CLINICAL TRIAL: NCT04092673
Title: A Phase 1-2 Dose-Escalation and Cohort-Expansion Study of Intravenous Zotatifin (eFT226) in Subjects With Selected Advanced Solid Tumor Malignancies
Brief Title: Study of eFT226 in Subjects With Selected Advanced Solid Tumor Malignancies
Acronym: Zotatifin
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Effector Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: eFT226-0002
Record Dates: First submitted 2019-09-10; First posted 2019-09-17 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — sotorasib; Fulvestrant; abemaciclib; Trastuzumab

STUDY DESIGN:
Intervention Model Description: Dose Escalation, 3+3, 3+3+3
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1: Sequential escalation (Completed) (Experimental): eFT226 administered IV weekly in 21-day cycles; dose escalated in sequential cohorts after subjects enrolled in a given cohort have completed DLT evaluation period.
  Interventions: Drug: eFT226
- Part 2: Cohort Expansion, Monotherapy, NSCLC, KRAS (EMNK) (Experimental): Cohort EMNK
  Interventions: Drug: eFT226
- Part 2: Cohort Expansion, Monotherapy, Breast, FGFR (EMBF) (Experimental): Cohort EMBF
  Interventions: Drug: eFT226
- Part 2: Cohort Expansion, Monotherapy, Breast, HER2 (EMBH) (Experimental): Cohort EMBH
  Interventions: Drug: eFT226
- Part 2: Cohort Expansion, Combination, Breast, Fulvestrant (ECBF) (Experimental): Cohort ECBF; Combination therapy partner administered per SOC at the approved dose.
  Interventions: Drug: Fulvestrant
- Part 2: Cohort Expansion, Combination, NSCLC, Sotorasib (ECNS) (Experimental): Cohort ECNS; Combination therapy partner administered per SOC at the approved dose.
  Interventions: Drug: Sotorasib
- Part 2: Cohort Expansion, Combination, Breast, Fulvestrant+Abemaciclib (ECBF+A) (Experimental): Cohort ECBF+A; Combination therapy partner administered per SOC at the approved dose.
  Interventions: Drug: Fulvestrant; Drug: Abemaciclib
- Part 2: Cohort Expansion, Combination, Breast, Trastuzumab (ECBT) (Experimental): Cohort ECBT; Combination therapy partner administered per SOC at the approved dose.
  Interventions: Drug: Trastuzumab
- Part 1a: Dose Escalation, Combination, Breast (Experimental): eFT226 administered IV weekly in 21-day cycles. Fulvestrant will also be given. Dose escalations per protocol.
  Interventions: Drug: Fulvestrant
- Part 1b Dose Escalation, Combination, Breast (Experimental): eFT226 administered IV every other week in 14-day cycles. Fulvestrant will also be given. Dose escalations per protocol.
  Interventions: Drug: Fulvestrant
- Part 2 Cohort Expansion, Combination, Breast, Fulvestrant, Cyclin D1 (Experimental): ECBF-D1; Combination therapy partner administered per SOC at the approved dose.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: eFT226 — eFT226 is a novel small-molecule, investigational drug being developed by eFFECTOR Therapeutics as an anticancer therapy. eFT226 is a potent and selective inhibitor of eIF4A1-mediated translation and selectively regulates the translation of a subset of mRNAs based on sequence specific recognition motifs in their 5'-UTR. eIF4A1 inhibition by eFT226 downregulates expression of receptor tyrosine kinases and KRAS, leading to decreased signaling through the PI3K/AKT and MAPK pathways. Preclinical efficacy testing of eFT226 demonstrates activity across models of solid tumor cancers with amplifications in HER2, FGFR1/2 and mutations in KRAS (including breast, NSCLC and CRC).
  Other Names: Selective translation inhibitor
  Arms: Part 1: Sequential escalation (Completed); Part 2: Cohort Expansion, Monotherapy, Breast, FGFR (EMBF); Part 2: Cohort Expansion, Monotherapy, Breast, HER2 (EMBH); Part 2: Cohort Expansion, Monotherapy, NSCLC, KRAS (EMNK)
Drug: Sotorasib — Recommended dosage: 960 mg orally once daily
  Other Names: Lumarkus
  Arms: Part 2: Cohort Expansion, Combination, NSCLC, Sotorasib (ECNS)
Drug: Fulvestrant — 500 mg administered intramuscularly on Days 1, 15, 29, and once monthly thereafter
  Other Names: Faslodex
  Arms: Part 1a: Dose Escalation, Combination, Breast; Part 1b Dose Escalation, Combination, Breast; Part 2 Cohort Expansion, Combination, Breast, Fulvestrant, Cyclin D1; Part 2: Cohort Expansion, Combination, Breast, Fulvestrant (ECBF); Part 2: Cohort Expansion, Combination, Breast, Fulvestrant+Abemaciclib (ECBF+A)
Drug: Abemaciclib — Dose in combination with fulvestrant: 150 mg twice daily
  Other Names: Verzenia
  Arms: Part 2: Cohort Expansion, Combination, Breast, Fulvestrant+Abemaciclib (ECBF+A)
Drug: Trastuzumab — 600 mg every 3 weeks
  Other Names: Herceptin
  Arms: Part 2: Cohort Expansion, Combination, Breast, Trastuzumab (ECBT)

SUMMARY:
This clinical trial is a Phase 1-2, open-label, sequential-group, dose-escalation and cohort-expansion study evaluating the safety, pharmacokinetics (PK), pharmacodynamics, and antitumor activity of Zotatifin (eFT226) in subjects with selected advanced solid tumor malignancies.

DETAILED DESCRIPTION:
Part 1 (Dose Escalation): Completed; Recommended Phase 2 Dose (RP2D) and Maximum Tolerated Dose (MTD) identified

Part 1a (Dose Escalation) This cohort will enroll patients with an advanced breast cancer that is refractory or intolerant to SOC therapy.

Part 1b (Dose Escalation) This cohort will enroll patients with an advanced breast cancer that is refractory or intolerant to SOC therapy.

Part 2 (Expansion Cohort) provides defined expansion cohorts to further explore the safety, pharmacology, and clinical activity of eFT226 monotherapy and in various combinations in subjects with previously treated advanced solid tumor malignancies.

ELIGIBILITY:
Key Criteria:

Parts 1a and 1b (Dose Escalation + Fulvestrant):

* Patient has histological or cytological confirmation of breast cancer.
* Patient has metastatic disease or locoregionally recurrent disease which is refractory or intolerant to existing therapy(ies) known to provide clinical benefit.
* Patient has had prior chemotherapy, endocrine therapy, or other therapy as follows:

  * Minimum of one prior line of therapy for advanced/metastatic disease.
  * Maximum of five prior lines of therapy for advanced/metastatic disease.
  * Recurrence or progression on at least one line of endocrine therapy in the advanced/metastatic disease setting.
  * Prior treatment has included a CDK4/6 inhibitor.
* Tumor is ER+ (defined as ER IHC staining > 0%).

Cohort EMNK:

* Patient has undergone treatment with platinum-based chemotherapy and an anti-PD-1/L1 agent, if appropriate.
* Tumor has a known KRAS-activating mutation; Patients with KRAS G12C mutations are excluded.

Cohort EMBF:

* Patient has had prior chemotherapy, endocrine therapy, or other therapy as follows:

  * Minimum of one prior line of therapy for advanced/metastatic disease.
  * Maximum of five prior lines of therapy for advanced/metastatic disease.
  * Recurrence or progression on at least one line of endocrine therapy in the advanced/metastatic disease setting, which may include combination therapy (eg, with a CDK4/6 inhibitor).
* Tumor is ER+ (defined as ER IHC staining > 0%) and has FGFR amplification.

Cohort EMBH:

* Patient has had prior chemotherapy, endocrine therapy, or other therapy as follows:

  * Minimum of one prior line of therapy for advanced/metastatic disease.
  * Minimum of one line of HER2-directed therapy Note: Prior treatment with CDK4/6 inhibitors is permitted.
* Tumor is ER+ (defined as ER IHC staining > 0%) and HER2+ (defined as HER2 3+ IHC staining or HER2 2+ and FISH+).

Cohort ECNS:

* Patient has histologically or cytologically confirmed stage IIIB (pleural or pericardial effusion) or stage IV NSCLC.
* Patient has undergone treatment with platinum-based chemotherapy and an anti-PD-1/L1 agent, if appropriate. Note: Patients who have declined approved therapy(ies) or who per treating physician are not eligible for approved therapy(ies) (eg, due to intolerance) may be eligible following discussion with the Medical Monitor.
* Tumor has a known G12C KRAS-activating mutation. Note: Patients who have been previously treated with KRAS-specific therapy are excluded.

Cohort ECBF:

* Patient has had prior chemotherapy, endocrine therapy, or other therapy as follows:

  * Minimum of one prior line of therapy for advanced/metastatic disease.
  * Maximum of five prior lines of therapy for advanced/metastatic disease.
  * Recurrence or progression on at least one line of endocrine therapy in the advanced/metastatic disease setting.
  * Prior treatment has included a CDK4/6 inhibitor.
* Tumor is ER+ (defined as ER IHC staining > 0%).

Cohort ECBF+A:

* Patient has had prior chemotherapy, endocrine therapy, or other therapy as follows:

  * Minimum of one prior line of therapy for advanced/metastatic disease.
  * Maximum of five prior lines of therapy for advanced/metastatic disease.
  * Recurrence or progression on at least one line of endocrine therapy in the advanced/metastatic disease setting.
* Tumor is ER+ (defined as ER IHC staining > 0%) and HER2- (defined as absence of HER2 3+ IHC staining and/or absence of FISH+).

Cohort ECBT:

* Patient has progressed after treatment with at least one approved anti-HER2 agent and has been administered at least one line of chemotherapy.
* Tumor is HER2+ (defined as HER2 3+ IHC staining or HER2 2+ and FISH+). Cohorts EMBF, EMBH, ECBF, ECBF+A: There is no limit on the number of lines of prior endocrine therapies.

Cohort ECBF-D1:

* Patient has metastatic disease or locoregionally recurrent disease which is refractory or intolerant to existing therapy(ies) known to provide clinical benefit.
* Patient has had prior chemotherapy, endocrine therapy, or other therapy as follows:

  * Minimum of one prior line of therapy for advanced/metastatic disease.
  * Maximum of five prior lines of therapy for advanced/metastatic disease.
  * Recurrence or progression on at least one line of endocrine therapy in the advanced/metastatic disease setting.
  * Prior treatment has included a CDK4/6 inhibitor.
* Tumor is ER+ (defined as ER IHC staining > 0%).
* Tumor has amplification of Cyclin D1 as determined by next generation sequencing or in situ hybridization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Parts 1a and 1b: MTD | Through study completion, approximately 12 months
  determined by occurrence of first cycle DLTs within a 3+3 or 3+3+3 clinical trial design
Parts 1a and 1b; incidence of AEs, serious adverse events (SAEs), and DLTs | Through study completion, approximately 12 months
  according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Parts 1a and 1b: RP2D | Through study completion, approximately 12 months
  determined by Incidence and type of DLTs
Parts 1a and 1b: RP2D | Through study completion, approximately 12 months
  determine by Incidence, type, and severity of AEs and SAEs graded as per NCI CTCAE
Part 2: Objective Response Rate- Efficacy | Through study completion, approximately 12 months
  defined as confirmed Complete Response (CR) or Partial Response (PR)
Part 2: (Combination Cohorts) Determine MTD | Through study completion, approximately 12 months
  determined by occurrence of first cycle Dose Limiting Toxicities (DLTs) within the study design
Part 2: (Combination Cohorts) Incidence, type, and severity of AEs and SAEs | Through study completion, approximately 12 months
  via adverse event monitoring
Part 2: (Combination Cohorts) Determine RP2D | Through study completion, approximately 12 months
  determined by incidence and type of DLTs, and incidence, type, and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Part 2: Percent change in tumor dimensions of target lesions- Efficacy | Through study completion, approximately 12 months
  calculated by the percentage change from baseline in the sum of the LD of target lesions
Part 2: Time to Response (TTR)- Efficacy | Through study completion, approximately 12 months
  defined as the interval from the start of study therapy to the first documentation of an objective response
Part 2: Duration of Response (DOR)- Efficacy | Through study completion, approximately 12 months
  defined as the interval from the first documentation of objective response to the earlier of the first documentation of disease progression or death from any cause

SECONDARY OUTCOMES:
Parts 1a and 1b: Objective response | Through study completion, approximately 12 months
  determined by confirmed CR or PR
Parts 1a and 1b: Percent change in tumor dimensions of target lesions | Through study completion, approximately 12 months
  calculated by the percentage change from baseline in the sum of the LD of target lesions
Parts 1a and 1b: TTR | Through study completion, approximately 12 months
  defined as the interval from the start of study therapy to the first documentation of an objective response
Parts 1a and 1b: DOR | Through study completion, approximately 12 months
  defined as the interval from the first documentation of objective response to the earlier of the first documentation of disease progression or death from any cause
Parts 1a and 1b: PFS | Through study completion, approximately 12 months
  defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression or death from any cause
Part 2: (Monotherapy and Combination Cohorts) Incidence and severity of AEs, SAEs, and additional safety parameters | Through study completion, approximately 12 months
  via adverse event monitoring
Part 2: Progression Free Survival | Through study completion, approximately 12 months
  defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression or death from any cause
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226 | Through study completion, approximately 12 months
  including area under the plasma concentration-time curve
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226 | Through study completion, approximately 12 months
  including maximum concentration
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226 | Through study completion, approximately 12 months
  including terminal phase rate constant
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226 | Through study completion, approximately 12 months
  including estimated steady-state volume of distribution [Vss]
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226 | Through study completion, approximately 12 months
  including half-life (t½)
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226 | Through study completion, approximately 12 months
  including total body clearance
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226including terminal state volume of distribution | Through study completion, approximately 12 months
  including terminal state volume of distribution
Evaluate plasma Pharmacokinetic (PK) parameters of eFT226 including terminal phase rate constant | Through study completion, approximately 12 months
  including terminal phase rate constant

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Warner, MD, Study Director — EFFECTOR Therapeutics, Inc.
Locations (14):
- United States (14):
  - University of Southern California, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University, Palo Alto, California
  - START Midwest, Grand Rapids, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center- Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center- Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center- Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center- David H. Koch Center for Cancer Care, New York, New York
  - University of Toledo Medical Center, Toledo, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - New Experimental Therapeutics of San Antonio - NEXT Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available